CLINICAL TRIAL: NCT05072613
Title: Pregnant Women Attending Antenatal Care Services as a Sentinel Population for Antimalarial Drug Resistance Genetic Surveillance in Africa
Brief Title: Monitoring Pregnant Women for Antimalarial Drug Resistance
Acronym: MIRANDA
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Kinshasa School of Public Health (Other); Wellcome Sanger Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 548-21
Record Dates: First submitted 2021-09-27; First posted 2021-10-11 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-05

CONDITIONS: Malaria
Keywords: Antimalarial Drug Resistance
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried Blood Spot. Only Plasmodium DNA will be analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: Pregnant women attending Antenatal Care Services
  Interventions: Other: Malaria screening
- School children: Children attending Primary Schools
  Interventions: Other: Malaria screening

INTERVENTIONS:
Other: Malaria screening — Participants are screened for malaria and a dried blood spot is collected from malaria positive cases

SUMMARY:
Annually, malaria affects an estimated 229 million people, causing 409,000 deaths (WHO 2019) mostly in Africa. Despite a substantial decline in malaria-related maternal and child deaths in recent years, progress in controlling malaria has been slower than anticipated and uneven across countries. COVID-19-related disruption of malaria control activities will likely further slow the pace and lead to an even greater burden in the near future.

One of the greatest challenges delaying progress in malaria elimination is antimalarial drug resistance. Recent reports of the emergence of artemisinin-resistant parasites in parts of Africa are the cause of even greater concern, since the loss of frontline treatment efficacy could bring about a dramatic reversal of progress.

Large-scale genetic surveillance of Plasmodium is an effective tool for rapid detection of changes in drug efficacy, enabling countries to switch to effective preventive and curative treatments when necessary. The implementation of genetic surveillance has proven very successful in small, low malaria burden countries. However, in large, high malaria burden countries such implementation is operationally and economically more complex.

Screening pregnant women attending Antenatal Care (ANC) services can be a practical and economical strategy for estimating malariometric parameters, with fewer limitations and challenges than conventional survey methodologies in children. The present study aims to demonstrate that this is also true for the genetic surveillance of antimalarial drug resistance.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy OR for children age <14 years old and in primary school

Exclusion Criteria:

* Refusal to participate (i.e., consent is not given by the participant for women or by the parents in the case of children)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women of all ages and in any trimester of pregnancy, and children <14 years old
Sampling Method: Non-Probability Sample
Enrollment: 6833 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Compare the frequency of Plasmodium falciparum mutations associated with antimalarial drug resistance in the population of pregnant women with that of children. | 18 months
  Plasmodium falciparum from infected individuals will be sequenced and the frequency of antimalarial drug resistance mutations in pregnant women will be compared with that of children.

SECONDARY OUTCOMES:
Evaluate the acceptability of the intervention | 12 months
  Acceptability will be measured as: 1) the number of women who agree to be tested for malaria, over the number of women who attend the ANC service and 2) via a specially designed questionnaire.
Compare malaria prevalence in pregnant women with that of in children throughout the year. | 12 months
  Malaria prevalence will be measured by Rapid Diagnostic Test and standard malaria microscopy in both populations (pregnant women and children) for a period of 12 months and results compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Kinshasa Medical Oxford Research Unit, Kinsasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunner NC, Chacky F, Mandike R, Mohamed A, Runge M, Thawer SG, Ross A, Vounatsou P, Lengeler C, Molteni F, Hetzel MW. The potential of pregnant women as a sentinel population for malaria surveillance. Malar J. 2019 Nov 21;18(1):370. doi: 10.1186/s12936-019-2999-0. PMID 31752889
- [Background] Mayor A, Menendez C, Walker PGT. Targeting Pregnant Women for Malaria Surveillance. Trends Parasitol. 2019 Sep;35(9):677-686. doi: 10.1016/j.pt.2019.07.005. Epub 2019 Aug 5. PMID 31395496
- [Background] van Eijk AM, Hill J, Noor AM, Snow RW, ter Kuile FO. Prevalence of malaria infection in pregnant women compared with children for tracking malaria transmission in sub-Saharan Africa: a systematic review and meta-analysis. Lancet Glob Health. 2015 Oct;3(10):e617-28. doi: 10.1016/S2214-109X(15)00049-2. Epub 2015 Aug 19. PMID 26296450
- [Background] Willilo RA, Molteni F, Mandike R, Mugalura FE, Mutafungwa A, Thadeo A, Benedictor E, Kafuko JM, Kaspar N, Ramsan MM, Mwaipape O, McElroy PD, Gutman J, Colaco R, Reithinger R, Ngondi JM. Pregnant women and infants as sentinel populations to monitor prevalence of malaria: results of pilot study in Lake Zone of Tanzania. Malar J. 2016 Jul 29;15(1):392. doi: 10.1186/s12936-016-1441-0. PMID 27473039
- [Derived] Onyamboko M, Wasakul V, Bakomba SB, Kayembe DK, Nzambiwishe BK, Ekombolo PE, Badjanga BB, Maindombe JM, Ngavuka JN, Lwadi BN, Drury E, Ariani C, Goncalves S, Chamsukhee V, Waithira N, Verschuuren TD, Lee SJ, Miotto O, Fanello C. Pregnant women as a sentinel population for genomic surveillance of malaria in the Democratic Republic of the Congo: a population-based study. Lancet Glob Health. 2025 Mar;13(3):e479-e487. doi: 10.1016/S2214-109X(24)00497-2. PMID 40021306